CLINICAL TRIAL: NCT01319721
Title: Limbal Conjunctival Autograft Versus Amniotic Membrane Graft When Combined With Mitomycin C for Recurrent Pterygium: A Randomized Trial
Brief Title: Recurrent Pterygium Surgery Using Mitomycin C With Limbal Conjunctival or Amniotic Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiyou Zhou (Other)
Responsible Party: Sponsor-Investigator, Shiyou Zhou, M.D., Ph.D., Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20101215
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Recurrent Pterygium
Keywords: Amniotic membrane; Limbal conjunctival autograft; Limbal; Conjunctival; Mitomycin C; Recurrent pterygium; Pterygium
MeSH Terms: conditions — Pterygium | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group LCAG (Active Comparator): After extensive excision of recurrent pterygium, intraoperative 0.2 mg/ml MMC (0.02%) for 3 minutes will be applied topically onto the exposed surgical area and then limbal conjunctival autograft for repairing the conjunctival defect.
  Interventions: Procedure: MMC; Procedure: AMG
- Group AMG (Active Comparator): After excision of recurrent pterygium, intraoperative 0.2 mg/ml MMC (0.02%) for 3 minutes will be applied topically onto the exposed surgical area and then an amniotic membrane graft for repairing the conjunctival defect.
  Interventions: Procedure: LCAG; Procedure: AMG

INTERVENTIONS:
Procedure: MMC — Intraoperative 0.2mg/ml mitomycin C (0.02%) for 3 minutes will be applied topically after extensive excision of recurrent pterygium.
  Other Names: mitomycin C
  Arms: Group LCAG
Procedure: LCAG — Limbal conjunctival autograft transplantation will be applied to closure of conjunctival defect after extensive excision of recurrent pterygium.
  Other Names: limbal conjunctiva; limbal conjunctival autograft; limbal conjunctival autograft transplantation
  Arms: Group AMG
Procedure: AMG — Amniotic membrane graft transplantation will be applied to closure of conjunctival defect after extensive excision of recurrent pterygium.
  Other Names: amniotic membrane graft; amniotic membrane transplantation; amniotic membrane graft transplantation

SUMMARY:
To compare the outcomes of limbal conjunctival autograft (LCAG) versus amniotic membrane graft (AMG) when combined with intraoperative 0.02% mitomycin C (MMC) after pterygium removal in patients with recurrent pterygium.

DETAILED DESCRIPTION:
Excision alone for treating recurrent pterygium was reported to be at risk of high recurrence again. As one of adjunctive methods, intraoperative application of a single dose of mitomycin C (MMC) seems to be the most commonly used method for preventing recurrence of pterygium. Additionally, closure of conjunctival defect after excision of pterygium by limbal conjunctival autograft or amniotic membrane have also become popular in recent years. There are a few reports in which MMC combined either limbal conjunctival autograft (LCAG) or amniotic membrane graft (AMG) for the treatment of recurrent pterygium. To assess the effectiveness and safety of these two combined approaches, the investigator plans to work on a randomized comparative and prospective trial of recurrent pterygium extensive excision with intraoperative 0.02% MMC application comparing LCAG to AMG.The patients enrolled in this study will be followed for at least 12 months after the surgery. Recurrence was defined as fibrovascular tissue crossing the limbus on to the clear cornea in the area of previous pterygium excision.

ELIGIBILITY:
Inclusion Criteria:

* The patients had one or two eye(s) with unilateral recurrent pterygium.
* Recurrent pterygium：be defined as of fibrovascular tissue onto the cornea for any distance in the position of a previous pterygium.
* Willingness to participate in research project and to attend research time.

Exclusion Criteria:

* Poor general health.
* Pregnant or lactating women.
* Patients with collagen vascular diseases or other autoimmune diseases.
* Patients with any evidence of stem cell deficiency.
* Patients with glaucoma who might require future filtering surgery.
* Patients with ocular infection.
* Patients with an allergy to mitomycin C, tobramycin or dexamethasone.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2010-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shiyou Zhou, MD, PHD, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- State Key Laboratory of Ophthalmology, Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients, who had one or two eye(s) with unilateral recurrent pterygium, were consecutively recruited from Zhongshan Ophthalmic Center, Guangzhou, between December 2010 and May 2013. In cases of bilateral eyes with recurrent pterygium, the left eye was the first to be assigned randomly, followed by the right eye.
Groups:
- Group LCAG: After excision of recurrent pterygium, intraoperative 0.2 mg/ml mitomycin C (0.02%) for 3 minutes will be applied topically onto the exposed surgical area and then limbal conjunctival autograft for repairing the conjunctival defect.
- Group AMG: After excision of recurrent pterygium, intraoperative 0.2 mg/ml mitomycin C (0.02%) for 3 minutes will be applied topically onto the exposed surgical area and then an amniotic membrane graft for repairing the conjunctival defect.
Period: Overall Study
Arm/Group | Group LCAG | Group AMG
Started | 48 (The unit of measure is eyes.) | 48 (The unit of measure is eyes.)
Completed | 47 (The unit of measure is eyes.) | 42 (The unit of measure is eyes.)
Not Completed | 1 | 6
Not completed — Lost to Follow-up | 1 | 6

BASELINE CHARACTERISTICS:
Population: No significant difference of the baseline characteristics was observed between the per-protocol population (n=89 eyes) and the randomized population (n=96 eyes), and there was no significant bias due to patients dropout. Therefore, the baseline participants for analysis were observed in the per-protocol population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group LCAG | Group AMG | Total
Number analyzed (Participants) | 47 | 42 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (12.2) | 55.3 (11.5) | 54.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 49
  Male | 20 | 20 | 40
Region of Enrollment [Number; unit: eyes]
  China | 47 | 42 | 89

OUTCOME MEASURES:

1. Primary Outcome: Recurrence
Description: Recurrence was defined as the presence of fibrovascular tissue in the surgical area and invasion onto the cornea. The appearance of the surgical bed in successful cases was graded as follows: grade A was defined as the operated eye being indistinguishable from a normal eye, grade B was defined as the presence of fine episcleral vessels without fibrous tissue in the surgical area extending up to the limbus but not beyond, and grade C was defined as the presence of fibrovascular tissue in the surgical area but without invasion onto the cornea.
Time Frame: One Year
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Group LCAG | Group AMG
Number analyzed (Participants) | 47 | 40
Number analyzed (eyes) | 47 | 42
eyes
  Grade A | 46 | 34
  Grade B | 0 | 3
  Grade C | 0 | 2
  Grade D (recurrence) | 1 | 3
Statistical Analysis 1: Comparison: Group LCAG vs Group AMG; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Complications
Time Frame: One year
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Group LCAG | Group AMG
Number analyzed (Participants) | 47 | 40
Number analyzed (eyes) | 47 | 42
eyes | 9 | 8
Statistical Analysis 1: Comparison: Group LCAG vs Group AMG; Test type: Superiority or Other; p < 0.05, Chi-squared

3. Secondary Outcome: Healing Time of Corneal Epithelial Defect
Time Frame: Four Weeks
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: eyes
Arm/Group | Group LCAG | Group AMG
Number analyzed (Participants) | 47 | 40
Number analyzed (eyes) | 47 | 42
days | 2.78 (0.73) | 3.25 (2.76)
Statistical Analysis 1: Comparison: Group LCAG vs Group AMG; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Eye Movement Amplitude (EMA)
Time Frame: One Year
Measure: Mean (Standard Deviation); unit: millimeter
Units Other Than Participants: eyes
Arm/Group | Group LCAG | Group AMG
Number analyzed (Participants) | 47 | 40
Number analyzed (eyes) | 47 | 42
millimeter
  Preoperative EMA | 6.67 (1.84) | 6.79 (2.01)
  Postoperative EMA | 8.35 (1.38) | 7.85 (1.94)
  Improvement of EMA | 1.67 (1.77) | 1.06 (1.84)
Statistical Analysis 1: Comparison: Group LCAG vs Group AMG; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

5. Secondary Outcome: Postoperative Conjunctival Inflammation
Description: The presence of conjunctival inflammation around the surgical site was assessed at 4 weeks post-operatively and graded as 0 (none), i (mild), ii (moderate), and iii (severe).
Time Frame: One month
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Group LCAG | Group AMG
Number analyzed (Participants) | 47 | 40
Number analyzed (eyes) | 47 | 42
eyes
  Grade 0 | 21 | 14
  Grade i | 17 | 14
  Grade ii | 9 | 13
  Grade iii | 0 | 1
Statistical Analysis 1: Comparison: Group LCAG vs Group AMG; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Group LCAG | Group AMG
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/40
Other Adverse Events (participants affected / at risk) | 9/47 | 7/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group LCAG (N=47) | Group AMG (N=40)
Punctate epithelial keratitis (Eye disorders) | 6 (6) | 5 (6)
Local episcleral melting (Eye disorders) | 2 (2) | 1 (1)
Localized pannus at donor site (Eye disorders) | 1 (1) | 0 (0)
Delayed epithelializaiton of corneal defect (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days